CLINICAL TRIAL: NCT02778139
Title: An Exploratory Study on the Risk Behaviours and Its Associated Psychosocial Factors in Hong Kong Chinese Youth Smokers
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Other Study IDs: UW 15-218
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Risk Behaviours

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- youth smokers
- non-smokers

SUMMARY:
The aims of this study were: (1) to examine the risk behaviours, lifestyle and its associated psychosocial factors for youth smokers; and (2) to explore the relationships among self-esteem, depressive symptoms and quality of life in youth smokers.

DETAILED DESCRIPTION:
The first approach is to conduct a qualitative interview on 30 youth smokers or until saturation, with the aim to examine the risk behaviours, lifestyle and its associated psychosocial factors for youth smokers.

Participants will be invited to complete a questionnaire on their demographic and socio-economic characteristics. An audiotaped semi-structured interview will then be conducted individually to each participant by two research assistants; with one research assistant will act as the interviewer to encourage the informants to freely express their feelings, thoughts and ideas and another will act as an observer and document any non-verbal language used by the informants. Prior to the data collection, written consent will be obtained from their parents and the participants will be invited to sign the child assent forms.

The second approach is to conduct a quantitative study to compare the self-esteem, depressive symptoms and quality of life between 100 youth smokers and 100 non-smokers.

For the quantitative approach, 100 youth smokers and 100 non-smokers will be recruited through the outreach programme organized by the smoking cessation research team of the School of Nursing. Such programme is a promotional activity to publicise the Youth Quitline and to raise the awareness of no smoking among youth in the community. A structured questionnaire will be used to obtain demographics and socio-economic characteristics of each subject.

Qualitative approach After completing the interviews, the recordings will be fully transcribed, verbatim, in Cantonese to capture nuances of expression unique to the dialect, and selected quotations relevant to the themes will be later translated into English. The analyses begin with an intensive examination of the transcriptions to search for general constructs and themes. Special attention will be given to constructs that diverged from the major topics as framed by the guiding questions.

The transcriptions will be first coded using the open coding method. As the number of codes grew, some closely related codes will be merged, resulting in a smaller, more manageable set of codes. Selective coding will then be adopted to code the transcriptions using the established categories. During the coding process, any inconsistencies in the interpretation of quotations or the assignment of codes will be resolved through discussions with the research team members. Finally, a complete set of codes will be generated to facilitate comparisons and the development of themes and categories.

Quantitative approach Data analysis will be performed using the SPSS, version 20.0 for Windows. The internal consistencies of various instruments used in the study will be determined by calculating their Cronbach. Descriptive statistics will be used to calculate the mean, standard deviation, and range of the scores of the different scales. The relationships among the scores of the CES-DC, RSES, PedsQL v. 4.0 and the participants' age, sex, education attainment, and smoking status will be investigated using the Pearson product-moment correlation coefficient. An independent t-test will be conducted to compare the mean scores of the CES-DC, RSES, PedsQL v. 4.0 between youth smokers and non-smokers.

ELIGIBILITY:
Inclusion Criteria:

* youth who are aged 25 or below
* smoke at least 1 cigarette in the past 30 days
* able to speak and understand Cantonese.

Exclusion Criteria:

* Have difficulty to communicate

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all current youth smokers aged 25 or below in Hong Kong
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The Centre for Epidemiologic Studies Depression Scale for Children (CES-DC) | baseline
  baseline depressive symptoms
The Rosenberg's Self-Esteem Scale (RSES) | baseline
  baseline self-esteem
Pediatric Quality-of-life Inventory (PedsQL v. 4.0) | baseline
  baseline quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Cheung Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: No